CLINICAL TRIAL: NCT03847922
Title: Nitrous Oxide for Analgesia During Office Urethral Bulking: a Randomized, Controlled Trial
Brief Title: Nitrous Oxide for Analgesia During Office Urethral Bulking
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to staffing changes in the hospital, we will be unable to complete this study for the requested 84 subjects. As such, we have decided to close this study.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 019-002
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2019-02

CONDITIONS: Pain; Stress Incontinence, Female
MeSH Terms: conditions — Pain; Urinary Incontinence, Stress | interventions — Nitrous Oxide; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with patients randomized 1:1 into two groups
Who Masked: Participant
Masking Description: Patients are blinded to their group assignment (they are not aware of whether they are receiving nitrous oxide or room air)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): lidocaine gel injected in the urethra 10 minutes prior to calcium hydroxylapatite injection plus self-administered room air
  Interventions: Drug: lidocaine gel 2%; Other: Room air
- Study group (Experimental): lidocaine gel injected in the urethra 10 minutes prior to calcium hydroxylapatite injection + self-administered Pro-Nox 50% nitrous oxide/50% oxygen.
  Interventions: Drug: Nitrous Oxide + Oxygen Gas (Product); Drug: lidocaine gel 2%

INTERVENTIONS:
Drug: Nitrous Oxide + Oxygen Gas (Product) — Self-administered 50% nitrous oxide / 50% oxygen mixture will be given to the intervention group, starting just before the beginning of the urethral bulking procedure.
  Other Names: Pro-Nox
  Arms: Study group
Drug: lidocaine gel 2% — 6mL of 2% lidocaine gel will be inserted and injected into the urethral canal approximately 10 minutes prior to the procedure for each participant regardless of group assignment.
  Other Names: Uro-Jet
Other: Room air — Room air will be administered via the Pro-Nox machine to participants in the control group, starting just before the beginning of the urethral bulking procedure.
  Arms: Control group

SUMMARY:
This study is designed to determine primarily if there is a difference in perceived pain in patients receiving urethral bulking with calcium hydroxylapatite using local lidocaine versus local lidocaine plus nitrous oxide gas. Patients will be randomized to a control group (local lidocaine plus room air) or a intervention group (local lidocaine plus 50% nitrous oxide/50% oxygen inhaled mixture). Their pain will be assessed immediately after the procedure, and their recollection of pain will also be assessed at their 2 week post-procedure visit. There are other secondary outcome measures as well; please see outcome measures section for full description.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* greater than or equal to 18 years old
* with demonstrable stress incontinence on supine stress test
* undergoing calcium hydroxylapatite injection for urethral bulking for the first time
* able to consent to the study and procedure

Exclusion Criteria:

* < 18 years old
* prior urethral bulking therapy
* predominant urge incontinence symptoms
* contraindications to nitrous oxide
* pre-existing significant cardiopulmonary disease
* hypotension defined as systolic blood pressure (BP) < 90 or diastolic BP <50 on initial BP in the office
* chronic pain disorders (specifically fibromyalgia, chronic pelvic pain, sciatica or chronic low back pain, painful bladder syndrome)
* chronic narcotic use (defined as taking a narcotic medication >3 days per week during the past two weeks)
* pregnancy
* conditions of air trapping (bullous emphysema, bowel obstruction, pneumothorax, intracranial air, middle ear conditions, status post recent diving, recent eye surgery)
* lidocaine allergy
* neurologic diseases impairing pain perception.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Change in pain | upon enrollment and immediately after the procedure
  Pain will be assessed both before the procedure upon enrollment immediately after the procedure using a 10cm visual analog scale (VAS), where patients will mark their pain level along the scale from "no pain" at 0cm to "pain as bad as it possibly could be" at 10cm; the change in pain score between the before and after procedure VASs (i.e. the baseline pain score subtracted from the post-procedure pain score) is the primary outcome

SECONDARY OUTCOMES:
Recollection of change in pain | 10 minutes after the procedure
  Recollection of pain measured by a 10cm visual analog scale (VAS) completed 10 minutes after the procedure; this will be compared to the baseline pain score on VAS from prior to the procedure, again to determine the patient's perceived change in pain during the procedure. The VAS used has patients mark their pain level along the scale from "no pain" at 0cm to "pain as bad as it possibly could be" at 10cm. The score on the VAS at baseline is subtracted from the score on the VAS at 10 minutes to get the change in pain as the patient remembered it.
Procedure time | Intra-procedure
  Time from the initial insertion of the cystoscope (for the injection of calcium hydroxylapatite) to final removal of the cystoscope
Change in Urogenital Distress Inventory (UDI-6) score | at enrollment and then again at the patient's 1-2 week post-procedure visit.
  A change in the patient's UDI-6 score, measured prior to procedure and then again at the 1-2 week post-procedure visit. UDI-6 is a measure of the severity of urinary symptoms the patient experiences, with minimum score of 0 (indicating no bother from urinary symptoms) and maximum score of 100 (indicating maximum bother from urinary symptoms). We will be assessing the change in this score from baseline, by subtracting the post-procedure score at 1-2 weeks from the baseline score.
Change in Incontinence Severity Index (ISI) score | at enrollment and then again at the patient's 1-2 week post-procedure visit.
  A change in the patient's ISI score, measured prior to procedure and then again at the 1-2 week post-procedure visit. ISI score measures severity of incontinence symptoms on a scale of 0 to 12, where 0 is no symptoms and 12 is maximal incontinence symptoms. We will calculate the change in score by subtracting the post-procedure score at 1-2 weeks from the baseline score.
Patient Global Impression of Improvement (PGI-I) score | 1-2 week post op visit
  Score on PGI-I at the patient's 1-2 week post-procedure visit. This score assesses who the patient feels their post-procedure condition is compared to prior to the procedure on a scale of 1-7, where 1 is "very much better" and 7 is "very much worse."
Adverse events | during the procedure
  apneic episodes > 15 seconds, patient lack of responsiveness, patient dissociative behavior, hypotension with blood pressure < 90/50, bradycardia < 50bpm, hypoxia with oxygen saturation <92% on pulse oximetry, significant nausea or vomiting
Blood pressure | during the procedure
  We will record blood pressure every 5 minutes during the procedure
Episodes of hypoxia | during the procedure
  We will record any oxygen saturation < 92% during the procedure
Episodes of bradycardia | during the procedure
  We will record any episodes of heart rate < 60bpm during the procedure
Episodes of tachycardia | during the procedure
  We will record episodes of heart rate > 100bpm during the procedure
Patient's suspected group assignment | 10 minutes after the procedure
  10 minutes after the procedure, the patients will be asked to which treatment arm they suspected they were allocated

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Hines, MD, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor Scott and White Medical Center, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Once all data is collected for a specific patient, it will be deidentified and entered in a spread sheet to be used for this study only.